CLINICAL TRIAL: NCT04304157
Title: A Prospective, Double Masked, up and Down Sequential Method to Estimate the Median Effective Dose of Dexmedetomidine in Elective Upper Limb Lidocaine Intravenous Regional Anesthesia
Brief Title: Median Effective Dose of Dexmedetomidine in Elective Upper Limb Lidocaine Intravenous Regional Anesthesia
Acronym: dexdix
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: South Valley University (Other)
Collaborators: Tanta University (Other)
Responsible Party: Principal Investigator, Ossama Hamdy Salman, Dr., South Valley University
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ossamahamdyresearch5
Record Dates: First submitted 2020-03-02; First posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Intravenous Drug Usage
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- satisfactory (Experimental): 0.4 µg.kg of dexmedetomidine, with 0.1 µg.kg dose interval. If IVRA outcome was satisfactory, the dose went down for the next patient by 0.1 µg.kg. Vice versa, if the outcome was unsatisfactory, the dexmedetomidine dose was stepped up by 0.1 µg.kg for the following patient
  Interventions: Drug: Dexmedetomidine
- unsatisfactory (Experimental): 0.4 µg.kg of dexmedetomidine, with 0.1 µg.kg dose interval. If IVRA outcome was satisfactory, the dose went down for the next patient by 0.1 µg.kg. Vice versa, if the outcome was unsatisfactory, the dexmedetomidine dose was stepped up by 0.1 µg.kg for the following patient
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine (DEX) a potent α 2 agonist that have unique analgesic, anxiolytic and sedative profile has been called upon as attractive adjunct in general as well as regional anesthesia with enticing results. Several studies have pursued DEX median effective dose (ED50) in different settings e.g., co induction agent with Propofol, in laryngeal muscle insertion and with local anesthetic to enhance the quality of spinal anesthesia
  Other Names: dixon's sequential method

SUMMARY:
Auxiliary drugs augment the effect of local anesthetic in intravenous regional anesthesia (IVRA). The purpose of our study was to estimate the median effective dose (ED50) of Dexmedetomidine in elective upper limb Lidocaine 0.5% IVRA.

DETAILED DESCRIPTION:
Since its innovation in 1908 by Dr August Bier of Germany, Intravenous regional anesthesia (IVRA) has stood the test of time as simple, safe and effective technique of regional anesthesia. 1 The technique entails insertion of intravenous catheter into a surgical limb before isolating it from the general circulation by tourniquet then inject local anesthetic (LA) into this isolated limb. 2 IVRA block is preferably used with short surgical procedures or maneuvers of the upper or lower extremity. Nevertheless, the technique has gained popularity for procedures of the upper extremity because of tourniquet issues like tourniquet pain, and other safety concerns that arise more often with lower extremity IVRA, essentially leakage of the of LA.3 Unfortunately, using LA solely for IVRA has not achieved optimum intraoperative analgesia or overcome the frequently reported tourniquet pain.4 A long list of adjuvants, to mention few: morphine, muscle relaxant and clonidine, have been used to augment LA action and ameliorate tourniquet pain. 5 Dexmedetomidine (DEX) a potent α 2 agonist that have unique analgesic, anxiolytic and sedative profile has been called upon as attractive adjunct in general as well as regional anesthesia with enticing results. Several studies have pursued DEX median effective dose (ED50) in different settings e.g., co induction agent with Propofol, in laryngeal muscle insertion and with local anesthetic to enhance the quality of spinal anesthesia. 6 However, DEX effective median dose ED50 with IVRA for upper limb has not been investigated elsewhere, so far. The up and down sequential method of Dixon and Mood is a common sequential design method used in anesthesia research to detect the ED50. It is a sequence of experiments performed under the assumption that "satisfactory response" is followed by decrease in test dose for the next patient in the series, and "non- satisfactory response" is followed by increase in test dose for the next patient in the series. 7 The purpose of this study is to estimate the median effective dose of Dexmedetomidine (DEX) with Lidocaine 0.5% IVRA in upper limb elective surgeries, using modified Dixon's up and down method.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 60 years
* American Society of Anesthesiologists physical status I or II
* Undergoing minor upper limb orthopedic surgical procedures in the hand, wrist and forearms including: metacarpal fracture, tendon injury, and carpal tunnel release.

Exclusion Criteria:

* Allergy to test drugs.
* vascular disease.
* contraindication to tourniquet applications.
* difficulty to manipulate the surgical limb.
* surgery expected to last more than an hour.
* patient refusal

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
1. Pain intensity measure | 8 hours
  Patients reported pain intensity at baseline, every 5 minutes during the surgery and every hour for 6 hours after the surgery. Pain intensity scored 0-10 (0 being no pain at all, and 10 the worst pain ever).

SECONDARY OUTCOMES:
Changes in mean blood pressure in mmHg | 8 h ours
  mean blood pressure in mmHg was measured at baseline, every 5 minutes during the surgery and every hour for 6 hours after the surgery
changes in heart rate (beat per minute) | 8 hours
  Changes in heart at baseline, every 5 minutes during the surgery and every hour for 6 hours after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Gad s Gad, MD, Study Director — South Valley University
Locations (1):
- South Valley University, Qina, Egypt

IPD SHARING:
Plan to Share IPD: No